CLINICAL TRIAL: NCT03429543
Title: A Double-blind, Randomised, Placebo-controlled, Parallel Group Trial to Evaluate the Efficacy and Safety of Empagliflozin and Linagliptin Over 26 Weeks, With a Double-blind Active Treatment Safety Extension Period up to 52 Weeks, in Children and Adolescents With Type 2 Diabetes Mellitus
Brief Title: Diabetes Study of Linagliptin and Empagliflozin in Children and Adolescents (DINAMO)TM
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1218-0091; 2016-000669-21 (EudraCT Number)
Record Dates: First submitted 2018-02-06; First posted 2018-02-12 (Actual); Results first posted 2024-02-23 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Metformin; Insulin; Linagliptin; empagliflozin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Placebo - DINAMOᵀᴹ & DINAMOᵀᴹ Mono (Placebo Comparator): Patients treated with metformin and/or insulin or patients who do not tolerate metformin or treatment-naïve patients or patients who are not on active treatment took 1 film-coated tablet of either Linagliptin or Empagliflozin matched placebo once daily, until end of treatment.
  Interventions: Drug: Metformin; Drug: Insulin; Drug: Placebo
- Placebo - Linagliptin 5 mg - DINAMOᵀᴹ & DINAMOᵀᴹ Mono (Experimental): Patients treated with metformin and/or insulin or patients who do not tolerate metformin or treatment-naïve patients or patients who are not on active treatment took 1 film-coated tablet of either Linagliptin or Empagliflozin matched placebo once daily, until end of treatment.
  Interventions: Drug: Metformin; Drug: Insulin; Drug: Placebo; Drug: Linagliptin
- Placebo - Empagliflozin 10 mg - DINAMOᵀᴹ & DINAMOᵀᴹ Mono (Experimental): Patients treated with metformin and/or insulin or patients who do not tolerate metformin or treatment-naïve patients or patients who are not on active treatment took 1 film-coated tablet of either Linagliptin or Empagliflozin matched placebo once daily. At week 26, patients were re-randomised to receive 10 milligram (mg) empagliflozin, taken once daily, until end of treatment.
  Interventions: Drug: Metformin; Drug: Insulin; Drug: Placebo; Drug: Empagliflozin
- Placebo - Empagliflozin 25 mg - DINAMOᵀᴹ & DINAMOᵀᴹ Mono (Experimental): Patients treated with metformin and/or insulin or patients who do not tolerate metformin or treatment-naïve patients or patients who are not on active treatment took 1 film-coated tablet of either Linagliptin or Empagliflozin matched placebo once daily. At week 26, patients were re-randomised to receive 25 milligram (mg) empagliflozin, taken once daily, until end of treatment.
  Interventions: Drug: Metformin; Drug: Insulin; Drug: Placebo; Drug: Empagliflozin
- Linagliptin 5 mg - DINAMOᵀᴹ & DINAMOᵀᴹ Mono (Experimental): Patients treated with metformin and/or insulin or patients who do not tolerate metformin or treatment-naïve patients or patients who are not on active treatment took 1 film-coated tablet of 5 milligram (mg) Linagliptin once daily, until end of treatment.
  Interventions: Drug: Metformin; Drug: Insulin; Drug: Linagliptin
- Empagliflozin 10 mg - DINAMOᵀᴹ & DINAMOᵀᴹ Mono (Experimental): Patients treated with metformin and/or insulin or patients who do not tolerate metformin or treatment-naïve patients or patients who are not on active treatment took 1 film-coated tablet of 10 milligram (mg) Empagliflozin once daily, until Week 14. Responder patients were not re-randomised at week 14 and continued 10 mg empagliflozin, taken once daily, until end of treatment. Non responder patients were re-randomised at Week 14 to receive 10 mg empagliflozin, taken once daily, until end of treatment.
  Interventions: Drug: Metformin; Drug: Insulin; Drug: Empagliflozin
- Empagliflozin 10 mg - Empagliflozin 25 mg - DINAMOᵀᴹ & DINAMOᵀᴹ Mono (Experimental): Patients treated with metformin and/or insulin or patients who do not tolerate metformin or treatment-naïve patients or patients who are not on active treatment took 1 film-coated tablet of 10 milligram (mg) Empagliflozin once daily until Week 14. Non responder patients were re-randomised at Week 14 to receive 25 mg empagliflozin, taken once daily, until end of treatment.
  Interventions: Drug: Metformin; Drug: Insulin; Drug: Empagliflozin

INTERVENTIONS:
Drug: Metformin — At least 1000 mg/day or up to a maximal tolerated dose.
Drug: Insulin — Basal or multiple dose injection.
Drug: Placebo — 1 film-coated tablet of either Linagliptin or Empagliflozin matched placebo once daily.
  Arms: Placebo - DINAMOᵀᴹ & DINAMOᵀᴹ Mono; Placebo - Empagliflozin 10 mg - DINAMOᵀᴹ & DINAMOᵀᴹ Mono; Placebo - Empagliflozin 25 mg - DINAMOᵀᴹ & DINAMOᵀᴹ Mono; Placebo - Linagliptin 5 mg - DINAMOᵀᴹ & DINAMOᵀᴹ Mono
Drug: Linagliptin — 1 film-coated tablet Linagliptin once daily, until end of treatment.
  Other Names: Trajenta(R)
  Arms: Linagliptin 5 mg - DINAMOᵀᴹ & DINAMOᵀᴹ Mono; Placebo - Linagliptin 5 mg - DINAMOᵀᴹ & DINAMOᵀᴹ Mono
Drug: Empagliflozin — 1 film-coated tablet of Empagliflozin once daily, until end of treatment.
  Other Names: Jardiance(R)
  Arms: Empagliflozin 10 mg - DINAMOᵀᴹ & DINAMOᵀᴹ Mono; Empagliflozin 10 mg - Empagliflozin 25 mg - DINAMOᵀᴹ & DINAMOᵀᴹ Mono; Placebo - Empagliflozin 10 mg - DINAMOᵀᴹ & DINAMOᵀᴹ Mono; Placebo - Empagliflozin 25 mg - DINAMOᵀᴹ & DINAMOᵀᴹ Mono

SUMMARY:
The purpose of this research study is to evaluate the efficacy and safety of an empagliflozin dosing regimen and one dose of linagliptin in patients with type 2 diabetes who are aged 10 to below 18 years and are currently taking metformin, insulin or both drugs (DINAMO TM) or who are treatment naïve or not on active treatment after metformin withdrawal (DINAMO TM MONO) .

Empagliflozin and linagliptin are both approved for use in adult patients with type 2 diabetes. This study will assess how well empagliflozin and linagliptin work by finding out how these treatments affect blood glucose (sugar) levels compared to placebo (a pill that contains no active drug), in children and adolescents. Empagliflozin and linagliptin are considered investigational products in this study since while they have been approved for use in adults, they have not been approved for children and adolescents due to lack of clinical studies in this specific population.

Patients with type 2 diabetes have higher levels of blood glucose (sugar) than patients who do not have this disease. The high level of sugar in the blood can lead to serious short-term and long-term medical problems. The main goal of treating diabetic patients is to lower blood glucose to a normal level. Lowering and controlling blood glucose help prevent or delay complications of diabetes such as heart disease, kidney, eye and nerve diseases, and the possibility of amputation.

Empagliflozin is a drug that helps to reduce blood glucose (sugar) levels by causing glucose to be excreted in the urines.

Linagliptin works by increasing the production of insulin (a hormone that controls the level of blood glucose) after meals when blood glucose (sugar) levels are too high. This helps to lower blood sugar levels.

The subject will either receive one of the active study drugs or a placebo. This study will be double blind; this means that neither the subject, nor the study doctor will know which treatment the subject will receive.

Which treatment the subject receives is decided by a computer, purely by chance; this is called a "random assignment".

For this study, there will first be a screening visit, followed by a 2-week placebo run-in period (all subjects will take placebo once daily). This run-in period is designed to ensure subjects are able to take the study drugs as described in the study protocol. Thereafter there will be a 26-week treatment phase (week 1-week 26) and a 26-week safety extension period (week 27-week 52). Following this there will be a follow-up visit at week 55.

On Day 1 after the placebo run-in phase, the subject will be randomly assigned to receive one of the 3 treatments: empagliflozin 10 mg, linagliptin 5 mg or placebo in a blinded manner. This treatment will continue up to week 14. Then after week 14, the subject will be assigned to receive one of the following 4 treatments: empagliflozin 10 mg, empagliflozin 25 mg, linagliptin 5 mg or placebo in a blinded manner. The drugs assigned after week 14 will be the same drugs as on Day 1 but some subjects will receive a higher dose of empagliflozin.

After the completion of the 26-week treatment period, the subject will enter a 26-week safety extension period. The same active treatment that the subject had been assigned to at week 14 visit will be continued. Subjects assigned to placebo on Day 1 will be randomly assigned to receive one of the 3 active treatments: empagliflozin 10 mg, empagliflozin 25 mg or linagliptin 5 mg in a blinded manner. This safety extension period is primarily designed to provide additional information on how well empagliflozin and linagliptin are tolerated.

Following the treatment phases, there will be a follow-up visit at week 55

Intervention model description:

Eligible subjects with HbA1c of 6.5% to 10.5% at screening will be randomized in a 1:1:1 ratio to receive empagliflozin 10 mg, linagliptin 5 mg or placebo. HbA1c assessment will be performed at Week 12. All subjects with Week 12 HbA1c < 7% will remain on previously assigned randomized treatment. Subjects taking empagliflozin with Week 12 HbA1c >= 7% will be re-randomized in a 1:1 ratio to continue on the low dose treatment (empagliflozin 10 mg) or up-titrate to the high dose treatment (empagliflozin 25 mg). Subjects taking linagliptin or placebo with Week 12 HbA1c >= 7% will remain on previously assigned treatment. All subjects will get new medication kits dispensed at Week 14 to maintain the blinding.

At Week 26, all subjects previously assigned to placebo will be re-randomized in a 1:1:1: ratio to receive one of the active treatments: empagliflozin 10 mg, empagliflozin 25 mg or linagliptin 5 mg. All subjects will get new medication kits dispensed at Week 14 to maintain the blinding.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 10 to 17 years (inclusive) at the time of randomisation (Visit 2)
* Male and female patients
* Women of childbearing potential (WOCBP) must be ready and able to use highly effective methods of birth control per ICH M3 (R2) that result in a low failure rate of less than 1% per year when used consistently and correctly. A list of contraception methods meeting these criteria is provided in the patient's legal representative information sheet.
* Signed and dated written informed consent provided by the patient's parent(s) (or legal guardian) and patient's assent in accordance with ICH-GCP and local legislation prior to admission to the trial (informed assent will be sought according to the patient's age, level of maturity, competence and capacity)
* Documented diagnosis of T2DM at Visit 1A:

  * DINAMO TM: Documented diagnosis of T2DM for at least 8 weeks at Visit 1A
  * DINAMO TM Mono: Confirmation of T2DM at Visit 1A
* Insufficient glycaemic control as measured by the central laboratory at Visit 1A:

  * DINAMO TM: HbA1c ≥ 6.5% and ≤ 10.5%
  * DINAMO TM Mono: HbA1c ≥ 6.5% and ≤ 9.0%
* DINAMO TM: Patients treated with

  * diet and exercise plus metformin at a stable dose for 8 weeks prior to Visit 2 or not tolerating metformin (defined as patients who were on metformin treatment for at least 1 week and had to discontinue metformin due to metformin-related side effects as assessed by the investigator) AND/OR
  * diet and exercise plus stable basal or MDI insulin therapy,, defined as a weekly average variation of the basal insulin dose ≤ 0.1 IU/kg over 8 weeks prior to Visit 2. - DINAMOTM Mono: Drug-naïve patients or patients not on active treatment (including discontinuation of metformin due to intolerance [or previous discontinuation for other reasons] and/or discontinuation of insulin [insulin use must be 8 weeks or less] at investigator's discretion) prior to or at Visit 1A)
* BMI ≥ 85th percentile for age and sex according to WHO references at Visit 1B
* Non-fasting serum C-peptide levels ≥ 0.6 ng/ml as measured by the central laboratory at Visit 1A
* Compliance with trial medication intake must be between 75% and 125% during the open-label placebo run-in period
* Further inclusion criteria apply

Exclusion Criteria:

* Any history of acute metabolic decompensation such as diabetic ketoacidosis within 8 weeks prior to Visit 1A and up to randomisation (mild to moderate polyuria at the time of randomisation is acceptable)
* Diagnosis of monogenic diabetes (e.g. MODY)
* History of pancreatitis
* Diagnosis of metabolic bone disease
* Gastrointestinal disorders that might interfere with study drug absorption according to investigator assessment
* Secondary obesity as part of a syndrome (e.g. Prader-Willi syndrome)
* Any antidiabetic medication (with the exception of metformin and/or insulin background therapy) within 8 weeks prior to Visit 1A and until Visit 2
* Treatment with weight reduction medications (including anti-obesity drugs) within 3 months prior to Visit 1A and until Visit 2
* History of weight-loss surgery or current aggressive diet regimen (according to investigator assessment) at Visit 1A and until Visit 2
* Treatment with systemic corticosteroids for > 1 week within 4 weeks prior to Visit 1A and up to Visit 2 Inhaled or topical use of corticosteroids (e.g. for asthma/chronic obstructive pulmonary disease) is acceptable.
* Change in dose of thyroid hormones within 6 weeks prior to Visit 1A or planned change or initiation of such therapy before Visit 2
* Known hypersensitivity or allergy to the investigational products or their excipients
* Impaired renal function defined as estimated Glomerular Filtration Rate (eGFR) < 60 ml/min/1.73m² (according to Zappitelli formula) as measured by the central laboratory at Visit 1A
* Indication of liver disease defined by serum level of either alanine transaminase (ALT), aspartate transaminase (AST) or alkaline phosphatase above 3 fold upper limit of normal (ULN) at Visit 1A as measured by the central laboratory at Visit 1A
* History of belonephobia (needle phobia)
* Any documented active or suspected malignancy or history of malignancy within 5 years prior to Visit 1A, except appropriately treated basal cell carcinoma of the skin or in situ carcinoma of uterine cervix
* Blood dyscrasias or any disorders causing haemolysis or unstable red blood cells (e.g. malaria, babesiosis, haemolytic anaemia)
* Any other acute or chronic medical or psychiatric condition or laboratory abnormality that, based on investigator's judgement, would jeopardize patient safety during trial participation or would affect the study outcome
* Medical contraindications to metformin according to the local label (for patient on metformin background therapy)
* Patient not able or cannot be supported by his/her parent(s) or legal guardian to understand and comply with study requirements based on investigator's judgement
* Previous randomisation in this trial
* Currently enrolled in another investigational device or drug trial, or less than 30 days since ending another investigational device or drug trial(s), or receiving other investigational treatment(s)
* Chronic alcohol or drug abuse within 3 months prior to Visit 1A or any condition that, in the investigator's opinion, makes them an unreliable trial patient or unlikely to complete the trial
* Female patients who are pregnant, nursing, or who plan to become pregnant in the trial

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 175 (Actual)
Dates: Start 2018-03-20 (Actual); Primary Completion 2022-10-19 (Actual); Study Completion 2023-05-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (83):
- United States (44):
  - Phoenix Children's Hospital, Phoenix, Arizona
  - University of Arizona, Tucson, Arizona
  - CHOC Children's Hospital, Orange, California
  - Stanford University Medical Center, Palo Alto, California
  - Rady Children's Hospital - San Diego, San Diego, California
  - University of California San Francisco, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Yale University School of Medicine, New Haven, Connecticut
  - Oceane7 Clinical Research, Miami, Florida
  - Empire Clinical Research, LLC, Miami Lakes, Florida
  - Pediatric and Adult Research Center, Orlando, Florida
  - Nemours Clinic, Pensacola, Florida
  - University of South Florida, Tampa, Florida
  - AdventHealth Medical Group, Pediatric Diabetes and Endocrinology at Winter Park, Winter Park, Florida
  - Children's Center for Advanced Pediatrics, Atlanta, Georgia
  - Atlanta Center, Atlanta, Georgia
  - Columbus Regional Research Institute, Columbus, Georgia
  - Rocky Mountain Diabetes and Osteoporosis Center, Idaho Falls, Idaho
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Novak Center for Children's Health, Louisville, Kentucky
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Boston Children's Hospital, Boston, Massachusetts
  - Joslin Diabetes Center, Boston, Massachusetts
  - Integrative Biosciences Center, Detroit, Michigan
  - University Of Mississippi Medical Center, Jackson, Mississippi
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - UBMD Pediatrics, Buffalo, New York
  - New York University Langone Medical Center, New York, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - Advantage Clinical Trials, The Bronx, New York
  - The University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - University Hospitals of Cleveland, Cleveland, Ohio
  - University of Oklahoma, Oklahoma City, Oklahoma
  - University of Oklahoma, Tulsa, Oklahoma
  - Penn State College of Medicine, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Monument Health Rapid City Hospital, Inc., Rapid City, South Dakota
  - LifeDoc Research, PLLC, Memphis, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Office of Amir A. Hassan, MD, P.A., Houston, Texas
  - Saenz Medical Center, La Joya, Texas
  - Texas Diabetes Institute, San Antonio, Texas
  - University of Virginia Health System, Charlottesville, Virginia
  - Children's Hospital of Richmond at VCU, Richmond, Virginia
- Argentina (2):
  - Sanatorio Allende S.A., Nueva Córdoba
  - Hospital de Clínicas Pte. Dr. Nicolás Avellaneda, San Miguel de Tucumán
- Brazil (2):
  - Instituto de Estudos e Pesquisas Clínicas IEP-CE, Fortaleza
  - Fundacao de Apoio ao Ensino, Pesquisa e Assistencia do Hospital das Clinicas da Faculdade de Medicina de Ribeirao Preto, Ribeirão Preto
- Canada (2):
  - University of Manitoba - Health Sciences Centre, Winnipeg, Manitoba
  - The Hospital for Sick Children, Toronto, Ontario
- China (2):
  - The First Hospital of Jilin University, Changchun
  - Zhengzhou Children'S Hospital, Zhengzhou
- Colombia (2):
  - Centro de Diabetes Cardiovascular IPS, Barranquilla
  - Dexa-Diab IPS, Bogotá DC
- Universitätsklinikum Freiburg, Freiburg im Breisgau, Germany
- Israel (3):
  - Soroka Univ. Medical Center, Beersheba
  - Rambam Medical Center, Haifa
  - The Chaim Sheba Medical Center Tel HaShomer, Ramat Gan
- Mexico (6):
  - Investigación en Salud y Metabolismo S.C., Chihuahua City
  - Centro de Estudios de Investigación Metabólicos y Cardiovasculares, S.C., Ciudad Madero
  - CAIMED Investigacion en Salud, S.A. de C.V., Mexico City
  - Consultorio Medico, Puebla City
  - Investigacion Medica Sonora S.C., Sonora
  - Centro de Investigación Médica de Ocidente, S.C., Zapopan
- San Juan Bautista School of Medicine, Caguas, Puerto Rico
- Russia (11):
  - Regional Clinical Hospital 'The Badge of Honor Order', Irkutsk
  - Ivanovo Reg.Clin.Hosp., Ivanovo
  - Rep.childrens clin.hosp., Izhevsk
  - State Medical University, Kazan, Kazan'
  - Munic. Instit. of HC "Kirov clin. hosp.#7 n.a.V.I.Urlova", Kirov
  - Endocrinology Scientific Center, MoH and Social Development, Moscow
  - State Novosibirsk Regional Clinical Hospital, Novosibirsk
  - Fed. State Budget Educational Instit. of Higher Education "Rostov State Med. Univ." of MoH of RF, Rostov-on-Don
  - St. Petersburg State Pediatric University, Saint Petersburg
  - Siberian State Med.Uni,Faculty Therapy Dep.w/ Clin.Pharmacol, Tomsk
  - Bahkir state med. Univ. of the Ministry Polyclinic Pediatric, Ufa
- South Korea (3):
  - Severance Hospital, Seoul
  - Asan Medical Center, Seoul
  - Ajou University Hospital, Suwon
- Thailand (2):
  - Rajavithi Hospital, Bangkok
  - Srinagarind Hospital, Khon Kaen
- United Kingdom (2):
  - St George's Hospital, London
  - Royal Berkshire Hospital, Reading

IPD SHARING:
Plan to Share IPD: Yes
After the study is completed and the primary manuscript is accepted for publishing, researchers can use this following link https://www.mystudywindow.com/msw/datasharing to request access to the clinical study documents regarding this study, and upon a signed "Document Sharing Agreement".
  Also, Researchers can use the following link https://www.mystudywindow.com/msw/datasharing to find information in order to request access to the clinical study data, for this and other listed studies, after the submission of a research proposal and according to the terms outlined in the website.
  The data shared are the raw clinical study data sets.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After all regulatory activities are completed in the US and EU for the product and indication, and after the primary manuscript has been accepted for publication.
Access Criteria: For study documents - upon signing of a 'Document Sharing Agreement'. For study data - 1. after the submission and approval of the research proposal (checks will be performed by both the independent review panel and the sponsor, including checking that the planned analysis does not compete with sponsor's publication plan); 2. and upon signing of a 'Data Sharing Agreement'.
URL: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- [Derived] Laffel LM, Danne T, Klingensmith GJ, Tamborlane WV, Willi S, Zeitler P, Neubacher D, Marquard J; DINAMO Study Group. Efficacy and safety of the SGLT2 inhibitor empagliflozin versus placebo and the DPP-4 inhibitor linagliptin versus placebo in young people with type 2 diabetes (DINAMO): a multicentre, randomised, double-blind, parallel group, phase 3 trial. Lancet Diabetes Endocrinol. 2023 Mar;11(3):169-181. doi: 10.1016/S2213-8587(22)00387-4. Epub 2023 Feb 1. PMID 36738751
- See also: Related Info — https://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was a randomised, placebo-controlled, double-blind, and parallel group trial with 3 treatment arms (placebo, 5 mg linagliptin, 10 mg empagliflozin). The main trial DINAMOᵀᴹ consisted of patients treated with metformin and/or insulin or patients who do not tolerate metformin. The ancillary trial DINAMOᵀᴹ Mono consisted of treatment-naïve patients or patients not on active treatment.
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria. Subjects were not to be allocated to a treatment group if any of the entry criteria were violated.
Groups:
- Placebo - Linagliptin 5 mg - DINAMOᵀᴹ & DINAMOᵀᴹ Mono: Patients treated with metformin and/or insulin or patients who do not tolerate metformin or treatment-naïve patients or patients who are not on active treatment took 1 film-coated tablet of either Linagliptin or Empagliflozin matched placebo once daily. At week 26, patients were re-randomised to receive 5 milligram (mg) Linagliptin, taken once daily, until end of treatment.
- Empagliflozin 10 mg - Empagliflozin 25 mg - DINAMOᵀᴹ & DINAMOᵀᴹ Mono: Patients treated with metformin and/or insulin or patients who do not tolerate metformin or treatment-naïve patients or patients who are not on active treatment who started on 10 milligram (mg) empagliflozin, taken once daily, who did not respond at Week 12 and were re-randomised at week 14 to receive 25 mg empagliflozin, taken once daily, until end of treatment.
Period: Overall Study
Arm/Group | Placebo - DINAMOᵀᴹ & DINAMOᵀᴹ Mono | Placebo - Linagliptin 5 mg - DINAMOᵀᴹ & DINAMOᵀᴹ Mono | Placebo - Empagliflozin 10 mg - DINAMOᵀᴹ & DINAMOᵀᴹ Mono | Placebo - Empagliflozin 25 mg - DINAMOᵀᴹ & DINAMOᵀᴹ Mono | Linagliptin 5 mg - DINAMOᵀᴹ & DINAMOᵀᴹ Mono | Empagliflozin 10 mg - DINAMOᵀᴹ & DINAMOᵀᴹ Mono | Empagliflozin 10 mg - Empagliflozin 25 mg - DINAMOᵀᴹ & DINAMOᵀᴹ Mono
Started | 7 | 19 | 16 | 16 | 59 | 45 | 13
Treated | 7 | 19 | 16 | 16 | 58 | 45 | 13
Completed | 0 | 17 | 15 | 14 | 47 | 36 | 12
Not Completed | 7 | 2 | 1 | 2 | 12 | 9 | 1
Not completed — Adverse Event | 1 | 1 | 0 | 0 | 0 | 2 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 5 | 0 | 1 | 2 | 6 | 3 | 1
Not completed — Other reason than listed | 0 | 1 | 0 | 0 | 4 | 4 | 0
Not completed — Not treated | 0 | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The randomised set (RS) included all randomised patients, regardless whether they took trial medication
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo - DINAMOᵀᴹ & DINAMOᵀᴹ Mono | Placebo - Linagliptin 5 mg - DINAMOᵀᴹ & DINAMOᵀᴹ Mono | Placebo - Empagliflozin 10 mg - DINAMOᵀᴹ & DINAMOᵀᴹ Mono | Placebo - Empagliflozin 25 mg - DINAMOᵀᴹ & DINAMOᵀᴹ Mono | Linagliptin 5 mg - DINAMOᵀᴹ & DINAMOᵀᴹ Mono | Empagliflozin 10 mg - DINAMOᵀᴹ & DINAMOᵀᴹ Mono | Empagliflozin 10 mg - Empagliflozin 25 mg - DINAMOᵀᴹ & DINAMOᵀᴹ Mono | Total
Number analyzed (Participants) | 7 | 19 | 16 | 16 | 59 | 45 | 13 | 175
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.3 (1.4) | 14.3 (1.7) | 14.1 (2.2) | 14.8 (1.8) | 14.4 (2.1) | 14.6 (1.8) | 13.9 (2.2) | 14.4 (1.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 12 | 11 | 8 | 36 | 31 | 8 | 112
  Male | 1 | 7 | 5 | 8 | 23 | 14 | 5 | 63
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 10 | 5 | 7 | 24 | 12 | 6 | 65
  Not Hispanic or Latino | 6 | 9 | 11 | 9 | 35 | 33 | 7 | 110
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian/Alaska Native | 0 | 1 | 0 | 0 | 3 | 4 | 0 | 8
  Asian | 0 | 1 | 1 | 1 | 5 | 2 | 0 | 10
  Black/African American | 5 | 4 | 3 | 6 | 17 | 20 | 4 | 59
  Native Hawaiian or other Pacific Islander | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 3
  White | 1 | 13 | 10 | 9 | 28 | 17 | 7 | 85
  Other including mixed or missing race | 1 | 0 | 1 | 0 | 4 | 2 | 2 | 10
HbA1c [Mean (Standard Deviation); unit: percentage] — HbA1c percentage Population: The treated set (TS) included all patients treated with at least 1 dose of randomised trial medication.
  percentage
    number analyzed (Participants) | 7 | 19 | 16 | 16 | 58 | 45 | 13 | 174
    (all) | 7.40 (0.77) | 8.01 (1.42) | 8.00 (1.28) | 8.14 (1.17) | 7.98 (1.09) | 7.78 (1.33) | 8.24 (1.08) | 7.94 (1.20)

OUTCOME MEASURES:

1. Primary Outcome: Change in Glycated Haemoglobin (HbA1c) (%) From Baseline to the End of 26 Weeks - DINAMOᵀᴹ
Description: Adjusted means taken from the following three models, as pre-specified in the protocol:
  Treatment group 1 (TG1): [Placebo], [Linagliptin 5mg] and [Empagliflozin pooled] Treatment group 2 (TG2): [Placebo] and [Empagliflozin 10mg and 10+25mg] Treatment group 3 (TG3): [Placebo] and [Empagliflozin 10mg]
  ANCOVA with continuous covariate (baseline HbA1c) and categorical covariates (treatment & age). Effect of linagliptin and of empagliflozin was compared with placebo at an overall α of 0.05 (2-sided) using the Hochberg method to account for multiple testing.
  After having obtained statistically significant results for both hypotheses of the primary family of hypotheses (TG1), the secondary hypotheses were to compare the individual empagliflozin doses versus placebo (TG2 & TG3). ANCOVA utilized a weight of zero for patients who were not in the hypothesis test of interest, a value of 2 for re-randomised patients who were in the hypothesis test of interest and a value of 1 otherwise.
Time Frame: Baseline (Day 1) and week 26 of treatment.
Population: Patients treated with at least 1 dose of trial medication who had a baseline HbA1c measurement. All data as observed were included. Any data after start of rescue medication and any on- and post-treatment values were kept. As pre-specified in the Protocol, endpoint only includes the DINAMOᵀᴹ data, subjects randomized to Empagliflozin were grouped in pre-specified treatment analysis groups (TG1, TG2, TG3) for hypotheses testing, data was not analyzed per individual arm.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent change
Groups:
- Placebo - DINAMOᵀᴹ (TG1, TG2 & TG3): Patients treated with metformin and/or insulin or patients who do not tolerate metformin took 1 film-coated tablet of either Linagliptin or Empagliflozin matched placebo once daily.
- Linagliptin 5 mg - DINAMOᵀᴹ (TG1): Patients treated with metformin and/or insulin or patients who do not tolerate metformin took 1 film-coated tablet of 5 milligram (mg) Linagliptin once daily.
- Empagliflozin Pooled (10 mg and 25 mg) - DINAMOᵀᴹ (TG1): Patients treated with metformin and/or insulin or patients who do not tolerate metformin took 1 film-coated tablet of 10 milligram (mg) Empagliflozin once daily. Patients who did not achieve an HbA1c value <7% at Week 12, were re-randomised to receive either 10 mg or 25 mg empagliflozin in a 1:1 ratio, taken once daily, until end of treatment.
- Empagliflozin 10 mg - DINAMOᵀᴹ (TG3): Patients treated with metformin and/or insulin or patients who do not tolerate metformin took 1 film-coated tablet of 10 milligram (mg) Empagliflozin once daily.
- Empagliflozin 10 mg - DINAMOᵀᴹ & Empagliflozin 10 - 25 mg - DINAMOᵀᴹ (TG2): Patients treated with metformin and/or insulin or patients who did not tolerate metformin started on 10 mg empagliflozin, taken once daily, who did achieve an HbA1c value <7% at Week 12 continued with 10 mg empagliflozin thereafter, until end of treatment.
  And
  Patients who started on 10 mg empagliflozin, taken once daily, who did not achieve an HbA1c value <7% at Week 12 and were re-randomised at week 14 to receive 25 mg empagliflozin, taken once daily, until end of treatment.
Arm/Group | Placebo - DINAMOᵀᴹ (TG1, TG2 & TG3) | Linagliptin 5 mg - DINAMOᵀᴹ (TG1) | Empagliflozin Pooled (10 mg and 25 mg) - DINAMOᵀᴹ (TG1) | Empagliflozin 10 mg - DINAMOᵀᴹ (TG3) | Empagliflozin 10 mg - DINAMOᵀᴹ & Empagliflozin 10 - 25 mg - DINAMOᵀᴹ (TG2)
Number analyzed (Participants) | 53 | 52 | 52 | 39 | 41
Percent change | NA [NA to NA] — TG1 Adjusted mean (95%CI): 0.68 (0.23, 1.13) TG2 Adjusted mean (95%CI): 0.66 (0.12, 1.21) TG3 Adjusted mean (95%CI): 0.68 (0.19, 1.17) | 0.33 [-0.13 to 0.79] | -0.17 [-0.64 to 0.31] | -0.49 [-1.03 to 0.04] | 0.14 [-0.42 to 0.71]
Statistical Analysis 1: Comparison: Placebo - DINAMOᵀᴹ (TG1, TG2 & TG3) vs Linagliptin 5 mg - DINAMOᵀᴹ (TG1); Treatment group 1 (TG1) consisting of Placebo, Linagliptin 5 mg and Empagliflozin pooled Patients: Analysis of covariance (ANCOVA) model with a continuous covariate (baseline HbA1c) and categorical covariates (treatment and age). The effect of linagliptin and of empagliflozin (including responders and non-responders) was compared with placebo at an overall α of 0.05 (2-sided) using the Hochberg method to account for multiple testing; Test type: Other; p = 0.2935, ANCOVA; Mean Difference (Final Values) = -0.34, 95% CI 2-sided [-0.99 to 0.30], Standard Error of Mean 0.33 — Mean difference calculated as [Treatment] - Placebo
Statistical Analysis 2: Comparison: Placebo - DINAMOᵀᴹ (TG1, TG2 & TG3) vs Empagliflozin Pooled (10 mg and 25 mg) - DINAMOᵀᴹ (TG1); [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.0116, ANCOVA; Mean Difference (Final Values) = -0.84, 95% CI 2-sided [-1.50 to -0.19], Standard Error of Mean 0.33 — Mean difference calculated as [Treatment] - Placebo
Statistical Analysis 3: Comparison: Placebo - DINAMOᵀᴹ (TG1, TG2 & TG3) vs Empagliflozin 10 mg - DINAMOᵀᴹ & Empagliflozin 10 - 25 mg - DINAMOᵀᴹ (TG2); Treatment group 2 (TG2) consisting of Placebo, Empagliflozin 25mg Patients: Analysis of covariance (ANCOVA) model with a continuous covariate (baseline HbA1c) and categorical covariates (treatment and age). The effect of linagliptin and of empagliflozin (including responders and non-responders) was compared with placebo at an overall α of 0.05 (2-sided) using the Hochberg method to account for multiple testing; Test type: Other — Only after having obtained statistically significant results for both hypotheses of the primary family of hypotheses (TG1), the secondary hypotheses were to compare the individual empagliflozin doses versus placebo based on TG2 and TG3.The ANCOVA utilised a weight of zero for patients who were not in the hypothesis test of interest, a value of 2 for re-randomised patients who were in the hypothesis test of interest and a value of 1 otherwise; p = 0.1943, ANCOVA; Mean Difference (Final Values) = -0.52, 95% CI 2-sided [-1.31 to 0.27], Standard Error of Mean 0.40 — Mean difference calculated as [Treatment] - Placebo
Statistical Analysis 4: Comparison: Placebo - DINAMOᵀᴹ (TG1, TG2 & TG3) vs Empagliflozin 10 mg - DINAMOᵀᴹ (TG3); Treatment group 3 (TG3) consisting of Placebo, Empagliflozin 10mg Patients: Analysis of covariance (ANCOVA) model with a continuous covariate (baseline HbA1c) and categorical covariates (treatment and age). The effect of linagliptin and of empagliflozin (including responders and non-responders) was compared with placebo at an overall α of 0.05 (2-sided) using the Hochberg method to account for multiple testing; Test type: Other — [test comment as in outcome 1, analysis 3]; p = 0.0015, ANCOVA; Mean Difference (Final Values) = -1.18, 95% CI 2-sided [-1.90 to -0.45], Standard Error of Mean 0.37 — Mean difference calculated as [Treatment] - Placebo

2. Primary Outcome: Percentage of Patients With Treatment Failure up to or at Week 26
Description: Percentage of patients with treatment failure up to or at Week 26 as a binary endpoint, defined as meeting at least one of the following criteria:
  * Use of rescue medication at any time up to Week 26
  * Increase from baseline in HbA1c by 0.5% at Week 26 . Increase from baseline in HbA1c to above 7.0% at Week 26 in patients with baseline HbA1c <7.0%
Time Frame: Up to 26 weeks.
Population: The modified intention-to-treat set (mITT) included all patients treated with at least 1 dose of trial medication who had a baseline HbA1c measurement. Missing values were regarded as 'treatment failures'. As pre-specified in the Protocol, endpoint only includes the ancillary study (DINAMOᵀᴹ Mono) data.
Measure: Number (90% Confidence Interval); unit: Percentage of subjects
Groups:
- Placebo - DINAMOᵀᴹ Mono: Treatment-naïve patients or patients who are not on active treatment took 1 film-coated tablet of either Linagliptin or Empagliflozin matched placebo once daily.
- Linagliptin 5 mg - DINAMOᵀᴹ Mono: Treatment-naïve patients or patients who are not on active treatment took 1 film-coated tablet of 5 milligram (mg) Linagliptin once daily.
- Empagliflozin Pooled (10 mg and 25 mg) - DINAMOᵀᴹ Mono: Treatment-naïve patients or patients who are not on active treatment took 1 film-coated tablet of 10 milligram (mg) Empagliflozin once daily. Patients who did not achieve an HbA₁c value <7% at Week 12, were re-randomised to receive either 10 mg or 25 mg empagliflozin in a 1:1 ratio, taken once daily, until end of treatment.
Arm/Group | Placebo - DINAMOᵀᴹ Mono | Linagliptin 5 mg - DINAMOᵀᴹ Mono | Empagliflozin Pooled (10 mg and 25 mg) - DINAMOᵀᴹ Mono
Number analyzed (Participants) | 5 | 6 | 6
Percentage of subjects | 60.0 [18.9 to 92.4] | 50.0 [15.3 to 84.7] | 50.0 [15.3 to 84.7]
Statistical Analysis 1: Comparison: Placebo - DINAMOᵀᴹ Mono vs Linagliptin 5 mg - DINAMOᵀᴹ Mono; Risk difference of active treatments versus placebo was determined and assessed by an exact 2-sided 90% confidence interval based on the method of Chan and Zhang. Patients were assigned to the treatment they were randomised to at the initial randomisation; Test type: Other; p = 1.0000, Fisher Exact; Risk Difference (RD) = -10.0, 90% CI 2-sided [-58.7 to 43.7] — Risk difference calculated as [treatment]-[placebo]
Statistical Analysis 2: Comparison: Placebo - DINAMOᵀᴹ Mono vs Empagliflozin Pooled (10 mg and 25 mg) - DINAMOᵀᴹ Mono; [analysis description as in outcome 2, analysis 1]; Test type: Other; p = 1.0000, Fisher Exact; Risk Difference (RD) = -10.0, 90% CI 2-sided [-58.7 to 43.7] — Risk difference calculated as [treatment]-[placebo]

3. Secondary Outcome: Change in HbA1c (%) From Baseline to the End of 26 Weeks - DINAMOᵀᴹ Mono
Description: Change in Glycated haemoglobin (HbA1c) (%) from baseline to the end of 26 weeks. Adjusted values came from a restricted maximum likelihood (REML) approach with mixed model for repeated measures (MMRM). Analyses included fixed categorical effects of treatment, visit, and treatment-by-visit interaction, as well as the categorical covariate age at randomisation and the continuous, fixed covariates of baseline of the response variable and baseline of the response variable-by-visit interaction. The covariate visit was treated as the repeated measure with an unstructured covariance structure used to model the within-patient measurements.
Time Frame: Baseline (Day 1) and week 26 of treatment.
Population: The modified intention-to-treat set (mITT) included all patients treated with at least 1 dose of trial medication who had a baseline HbA1c measurement. All available data as observed were included. Any values after start of rescue medication and any on- and post-treatment values were kept. As pre-specified in the Protocol, endpoint only includes the ancillary study (DINAMOᵀᴹ Mono) data.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent change
Groups:
- Placebo - DINAMOᵀᴹ Mono: Patients treated with metformin and/or insulin or patients who do not tolerate metformin took 1 film-coated tablet of either Linagliptin or Empagliflozin matched placebo once daily.
Arm/Group | Placebo - DINAMOᵀᴹ Mono | Linagliptin 5 mg - DINAMOᵀᴹ Mono | Empagliflozin Pooled (10 mg and 25 mg) - DINAMOᵀᴹ Mono
Number analyzed (Participants) | 4 | 5 | 4
Percent change | 0.15 [-1.45 to 1.75] | -0.53 [-2.01 to 0.95] | -0.23 [-1.83 to 1.37]
Statistical Analysis 1: Comparison: Placebo - DINAMOᵀᴹ Mono vs Linagliptin 5 mg - DINAMOᵀᴹ Mono; Restricted maximum likelihood (REML) approach with mixed model for repeated measures (MMRM). Fixed categorical effects of treatment, visit, and treatment-by-visit interaction and categorical covariate age (baseline) and continuous, fixed covariates of baseline of response variable and baseline of response variable-by-visit interaction. Covariate visit was treated as repeated measure with an unstructured covariance structure used to model within-patient measurements; Test type: Other; p = 0.4828, Mixed Models Analysis; Adjusted mean difference = -0.68, 95% CI 2-sided [-2.86 to 1.49] — Mean difference calculated as [Treatment] - Placebo
Statistical Analysis 2: Comparison: Placebo - DINAMOᵀᴹ Mono vs Empagliflozin Pooled (10 mg and 25 mg) - DINAMOᵀᴹ Mono; [analysis description as in outcome 3, analysis 1]; Test type: Other; p = 0.7047, Mixed Models Analysis; Adjusted mean difference = -0.38, 95% CI 2-sided [-2.64 to 1.88] — Mean difference calculated as [Treatment] - Placebo

4. Secondary Outcome: Time to Treatment Failure
Description: Time to treatment failure was analysed by Kaplan-Meier estimates up to the end of the study (Week 52). Patients in the placebo group were censored after 26 weeks unless a prior treatment failure was observed.
Time Frame: Up to 395 days.
Population: The modified intention-to-treat set (mITT) included all patients treated with at least 1 dose of trial medication who had a baseline HbA1c measurement. Missing values were regarded as 'failures'. As pre-specified in the Protocol, endpoint only includes the ancillary study (DINAMOᵀᴹ Mono) data.
Measure: Mean (Standard Error); unit: Days
Groups:
- Placebo - DINAMOᵀᴹ Mono: Treatment-naïve patients or patients who are not on active treatment took 1 film-coated tablet of either Linagliptin or Empagliflozin matched placebo once daily. At week 26, patients on placebo were re-randomised to receive either 5 mg linagliptin or 10 mg empagliflozin or 25 mg empagliflozin in a 1:1:1 ratio, taken once daily, until end of treatment.
- Linagliptin 5 mg - DINAMOᵀᴹ Mono: Patients treated with metformin and/or insulin or patients who do not tolerate metformin took 1 film-coated tablet of 5 milligram (mg) Linagliptin once daily.
- Empagliflozin Pooled (10 mg and 25 mg) - DINAMOᵀᴹ Mono: Patients treated with metformin and/or insulin or patients who do not tolerate metformin took 1 film-coated tablet of 10 milligram (mg) Empagliflozin once daily. Patients who did not achieve an HbA1c value <7% at Week 12, were re-randomised to receive either 10 mg or 25 mg empagliflozin in a 1:1 ratio, taken once daily, until end of treatment.
Arm/Group | Placebo - DINAMOᵀᴹ Mono | Linagliptin 5 mg - DINAMOᵀᴹ Mono | Empagliflozin Pooled (10 mg and 25 mg) - DINAMOᵀᴹ Mono
Number analyzed (Participants) | 5 | 6 | 6
Days | 65.600 (19.941) | 72.167 (20.280) | 167.333 (26.711)
Statistical Analysis 1: Comparison: Placebo - DINAMOᵀᴹ Mono vs Linagliptin 5 mg - DINAMOᵀᴹ Mono; Time to treatment failure was analysed by Kaplan-Meier estimates up to the end of the study. A log-rank test compared linagliptin and empagliflozin pooled versus placebo up to Week 26; Test type: Other; p = 0.8626, Log Rank
Statistical Analysis 2: Comparison: Placebo - DINAMOᵀᴹ Mono vs Empagliflozin Pooled (10 mg and 25 mg) - DINAMOᵀᴹ Mono; [analysis description as in outcome 4, analysis 1]; Test type: Other; p = 0.2827, Log Rank

5. Secondary Outcome: Change in Fasting Plasma Glucose (FPG, mg/dL) From Baseline to the End of 26 Weeks
Description: Change in fasting plasma glucose (FPG, Milligrams Per Deciliter (mg/dL)) from baseline to the end of 26 weeks. Adjusted values taken from analysis of covariance (ANCOVA) model with treatment as a fixed classification effect, baseline FPG as linear covariate and age at randomisation as categorical covariate. The random error was assumed to be normally distributed.
Time Frame: Baseline (Day 1) and week 26.
Population: The modified intention-to-treat set (mITT) included all patients treated with at least 1 dose of trial medication who had a baseline HbA1c measurement. All available data as observed were included. Any values after start of rescue medication and any on- and post-treatment values were kept, baseline observations were carried forward to impute the missing data. Only patients with non-missing data were included.
Measure: Least Squares Mean (95% Confidence Interval); unit: Milligrams Per Deciliter (mg/dL)
Groups:
- Placebo - DINAMOᵀᴹ: Patients treated with metformin and/or insulin or patients who do not tolerate metformin took 1 film-coated tablet of either Linagliptin or Empagliflozin matched placebo once daily.
- Linagliptin 5 mg - DINAMOᵀᴹ: Patients treated with metformin and/or insulin or patients who do not tolerate metformin took 1 film-coated tablet of 5 milligram (mg) Linagliptin once daily.
- Empagliflozin Pooled (10 mg and 25 mg) - DINAMOᵀᴹ: Patients treated with metformin and/or insulin or patients who do not tolerate metformin took 1 film-coated tablet of 10 milligram (mg) Empagliflozin once daily. Patients who did not achieve an HbA1c value <7% at Week 12, were re-randomised to receive either 10 mg or 25 mg empagliflozin in a 1:1 ratio, taken once daily, until end of treatment.
- Placebo - DINAMOᵀᴹ Mono: Patients treated with metformin and/or insulin or patients who do not tolerate metformin took 1 film-coated tablet of either Linagliptin or Empagliflozin matched placebo once daily. At week 26, patients on placebo were re-randomised to receive either 5 mg linagliptin or 10 mg empagliflozin or 25 mg empagliflozin in a 1:1:1 ratio, taken once daily, until end of treatment.
Arm/Group | Placebo - DINAMOᵀᴹ | Linagliptin 5 mg - DINAMOᵀᴹ | Empagliflozin Pooled (10 mg and 25 mg) - DINAMOᵀᴹ | Placebo - DINAMOᵀᴹ Mono | Linagliptin 5 mg - DINAMOᵀᴹ Mono | Empagliflozin Pooled (10 mg and 25 mg) - DINAMOᵀᴹ Mono
Number analyzed (Participants) | 52 | 51 | 48 | 4 | 4 | 5
Milligrams Per Deciliter (mg/dL) | 15.70 [-0.53 to 31.93] | 10.29 [-6.12 to 26.69] | -19.48 [-36.39 to -2.57] | -38.50 [-62.67 to -14.33] | 0.12 [-23.67 to 23.91] | -18.45 [-40.00 to 3.10]
Statistical Analysis 1: Comparison: Placebo - DINAMOᵀᴹ vs Linagliptin 5 mg - DINAMOᵀᴹ; Analysis of covariance (ANCOVA) model with treatment as a fixed classification effect, baseline FPG as linear covariate and age at randomisation as categorical covariate. The random error was assumed to be normally distributed; Test type: Other; p = 0.6438, ANCOVA; Mean Difference (Final Values) = -5.41, 95% CI 2-sided [-28.49 to 17.67] — Mean difference calculated as [Treatment] - Placebo
Statistical Analysis 2: Comparison: Placebo - DINAMOᵀᴹ vs Empagliflozin Pooled (10 mg and 25 mg) - DINAMOᵀᴹ; [analysis description as in outcome 5, analysis 1]; Test type: Other; p = 0.0035, ANCOVA; Mean Difference (Final Values) = -35.18, 95% CI 2-sided [-58.61 to -11.74] — Mean difference calculated as [Treatment] - Placebo
Statistical Analysis 3: Comparison: Placebo - DINAMOᵀᴹ Mono vs Linagliptin 5 mg - DINAMOᵀᴹ Mono; [analysis description as in outcome 5, analysis 1]; Test type: Other; p = 0.0310, ANCOVA; Mean Difference (Final Values) = 38.62, 95% CI 2-sided [4.54 to 72.70] — Mean difference calculated as [Treatment] - Placebo
Statistical Analysis 4: Comparison: Placebo - DINAMOᵀᴹ Mono vs Empagliflozin Pooled (10 mg and 25 mg) - DINAMOᵀᴹ Mono; [analysis description as in outcome 5, analysis 1]; Test type: Other; p = 0.1994, ANCOVA; Mean Difference (Final Values) = 20.05, 95% CI 2-sided [-13.01 to 53.11] — Mean difference calculated as [Treatment] - Placebo

6. Secondary Outcome: Change in Body Weight (kg) From Baseline to the End of 26 Weeks
Description: Change in body weight (kg) from baseline to the end of 26 weeks. Adjusted values taken from mixed model for repeated measures (MMRM) with the fixed categorical effects of treatment, visit, and treatment-by-visit interaction, as well as the categorical covariate age at randomisation and the continuous, fixed covariates of baseline of the response variable and baseline of the response variable-by-visit interaction. The covariate visit was treated as repeated measure with an unstructured covariance structure used to model the within-patient measurements.
Time Frame: Baseline (Day 1) and week 26.
Population: The modified intention-to-treat set (mITT) included all patients treated with at least 1 dose of trial medication who had a baseline HbA1c measurement. All available data as observed were included. Any values after start of rescue medication and any on- and post-treatment values were kept. Only patients with non-missing data were included.
Measure: Least Squares Mean (95% Confidence Interval); unit: kilogram (kg)
Groups:
- Empagliflozin Pooled (10 mg and 25 mg): Patients treated with metformin and/or insulin or patients who do not tolerate metformin took 1 film-coated tablet of 10 milligram (mg) Empagliflozin once daily. Patients who did not achieve an HbA1c value <7% at Week 12, were re-randomised to receive either 10 mg or 25 mg empagliflozin in a 1:1 ratio, taken once daily, until end of treatment.
Arm/Group | Placebo - DINAMOᵀᴹ | Linagliptin 5 mg - DINAMOᵀᴹ | Empagliflozin Pooled (10 mg and 25 mg) | Placebo - DINAMOᵀᴹ Mono | Linagliptin 5 mg - DINAMOᵀᴹ Mono | Empagliflozin Pooled (10 mg and 25 mg) - DINAMOᵀᴹ Mono
Number analyzed (Participants) | 50 | 49 | 48 | 4 | 6 | 4
kilogram (kg) | -0.04 [-1.40 to 1.32] | 1.42 [0.04 to 2.81] | -0.79 [-2.17 to 0.59] | 2.64 [-0.35 to 5.63] | 2.69 [0.24 to 5.14] | 1.29 [-1.75 to 4.33]
Statistical Analysis 1: Comparison: Placebo - DINAMOᵀᴹ vs Linagliptin 5 mg - DINAMOᵀᴹ; Mixed model for repeated measures (MMRM) with the fixed categorical effects of treatment, visit, and treatment-by-visit interaction, as well as the categorical covariate age at randomisation and the continuous, fixed covariates of baseline of the response variable and baseline of the response variable-by-visit interaction. The covariate visit was treated as repeated measure with an unstructured covariance structure used to model the within-patient measurements; Test type: Other; p = 0.1394, Mixed Models Analysis; Mean Difference (Final Values) = 1.46, 95% CI 2-sided [-0.48 to 3.41] — Mean difference calculated as [Treatment] - Placebo
Statistical Analysis 2: Comparison: Placebo - DINAMOᵀᴹ vs Empagliflozin Pooled (10 mg and 25 mg); [analysis description as in outcome 6, analysis 1]; Test type: Other; p = 0.4476, Mixed Models Analysis; Mean Difference (Final Values) = -0.75, 95% CI 2-sided [-2.68 to 1.19] — Mean difference calculated as [Treatment] - Placebo
Statistical Analysis 3: Comparison: Placebo - DINAMOᵀᴹ Mono vs Linagliptin 5 mg - DINAMOᵀᴹ Mono; [analysis description as in outcome 6, analysis 1]; Test type: Other; p = 0.9789, Mixed Models Analysis; Mean Difference (Final Values) = 0.05, 95% CI 2-sided [-3.80 to 3.90] — Mean difference calculated as [Treatment] - Placebo
Statistical Analysis 4: Comparison: Placebo - DINAMOᵀᴹ Mono vs Empagliflozin Pooled (10 mg and 25 mg) - DINAMOᵀᴹ Mono; [analysis description as in outcome 6, analysis 1]; Test type: Other; p = 0.5092, Mixed Models Analysis; Mean Difference (Final Values) = -1.35, 95% CI 2-sided [-5.68 to 2.99] — Mean difference calculated as [Treatment] - Placebo

7. Secondary Outcome: Change in Systolic Blood Pressure (SBP, mmHg) From Baseline to the End of 26 Weeks
Description: Change in systolic blood pressure (SBP, millimeters of mercury (mmHg)) from baseline to the end of 26 weeks. Adjusted values taken from mixed model for repeated measures (MMRM) with the fixed categorical effects of treatment, visit, and treatment-by-visit interaction, as well as the categorical covariate age at randomisation and the continuous, fixed covariates of baseline of the response variable and baseline of the response variable-by-visit interaction. The covariate visit was treated as repeated measure with an unstructured covariance structure used to model the within-patient measurements.
Time Frame: Baseline (Day 1) and week 26.
Population: as for outcome 6
Measure: Least Squares Mean (95% Confidence Interval); unit: millimeters of mercury (mmHg)
Arm/Group | Placebo - DINAMOᵀᴹ | Linagliptin 5 mg - DINAMOᵀᴹ | Empagliflozin Pooled (10 mg and 25 mg) - DINAMOᵀᴹ | Placebo - DINAMOᵀᴹ Mono | Linagliptin 5 mg - DINAMOᵀᴹ Mono | Empagliflozin Pooled (10 mg and 25 mg) - DINAMOᵀᴹ Mono
Number analyzed (Participants) | 50 | 49 | 48 | 4 | 6 | 4
millimeters of mercury (mmHg) | 1.30 [-1.01 to 3.61] | 2.21 [-0.14 to 4.56] | -0.12 [-2.47 to 2.24] | 2.63 [-4.07 to 9.34] | 5.16 [-0.74 to 11.06] | 2.63 [-4.86 to 10.12]
Statistical Analysis 1: Comparison: Placebo - DINAMOᵀᴹ vs Linagliptin 5 mg - DINAMOᵀᴹ; [analysis description as in outcome 6, analysis 1]; Test type: Other; p = 0.5870, Mixed Models Analysis; Mean Difference (Final Values) = 0.91, 95% CI 2-sided [-2.40 to 4.22] — Mean difference calculated as [Treatment] - Placebo
Statistical Analysis 2: Comparison: Placebo - DINAMOᵀᴹ vs Empagliflozin Pooled (10 mg and 25 mg) - DINAMOᵀᴹ; [analysis description as in outcome 6, analysis 1]; Test type: Other; p = 0.3967, Mixed Models Analysis; Mean Difference (Final Values) = -1.42, 95% CI 2-sided [-4.72 to 1.88] — Mean difference calculated as [Treatment] - Placebo
Statistical Analysis 3: Comparison: Placebo - DINAMOᵀᴹ Mono vs Linagliptin 5 mg - DINAMOᵀᴹ Mono; [analysis description as in outcome 6, analysis 1]; Test type: Other; p = 0.5414, Mixed Models Analysis; Mean Difference (Final Values) = 2.53, 95% CI 2-sided [-6.42 to 11.47] — Mean difference calculated as [Treatment] - Placebo
Statistical Analysis 4: Comparison: Placebo - DINAMOᵀᴹ Mono vs Empagliflozin Pooled (10 mg and 25 mg) - DINAMOᵀᴹ Mono; [analysis description as in outcome 6, analysis 1]; Test type: Other; p = 0.9995, Mixed Models Analysis; Mean Difference (Final Values) = 0.00, 95% CI 2-sided [-10.13 to 10.13] — Mean difference calculated as [Treatment] - Placebo

8. Secondary Outcome: Change in Diastolic Blood Pressure (DBP, mmHg) From Baseline to the End of 26 Weeks
Description: Change in diastolic blood pressure (DBP, millimeters of mercury (mmHg)) from baseline to the end of 26 weeks. Adjusted values taken from mixed model for repeated measures (MMRM) with the fixed categorical effects of treatment, visit, and treatment-by-visit interaction, as well as the categorical covariate age at randomisation and the continuous, fixed covariates of baseline of the response variable and baseline of the response variable-by-visit interaction. The covariate visit was treated as repeated measure with an unstructured covariance structure used to model the within-patient measurements.
Time Frame: Baseline (Day 1) and week 26.
Population: as for outcome 6
Measure: Least Squares Mean (95% Confidence Interval); unit: millimeters of mercury (mmHg)
Arm/Group | Placebo - DINAMOᵀᴹ | Linagliptin 5 mg - DINAMOᵀᴹ | Empagliflozin Pooled (10 mg and 25 mg) - DINAMOᵀᴹ | Placebo - DINAMOᵀᴹ Mono | Linagliptin 5 mg - DINAMOᵀᴹ Mono | Empagliflozin Pooled (10 mg and 25 mg) - DINAMOᵀᴹ Mono
Number analyzed (Participants) | 50 | 49 | 48 | 4 | 6 | 4
millimeters of mercury (mmHg) | 0.76 [-1.01 to 2.53] | 2.26 [0.46 to 4.05] | 0.78 [-1.04 to 2.60] | 3.42 [-4.92 to 11.75] | 6.75 [0.14 to 13.35] | -3.20 [-10.10 to 3.69]
Statistical Analysis 1: Comparison: Placebo - DINAMOᵀᴹ vs Linagliptin 5 mg - DINAMOᵀᴹ; [analysis description as in outcome 6, analysis 1]; Test type: Other; p = 0.2433, Mixed Models Analysis; Mean Difference (Final Values) = 1.50, 95% CI 2-sided [-1.03 to 4.02] — Mean difference calculated as [Treatment] - Placebo
Statistical Analysis 2: Comparison: Placebo - DINAMOᵀᴹ vs Empagliflozin Pooled (10 mg and 25 mg) - DINAMOᵀᴹ; [analysis description as in outcome 6, analysis 1]; Test type: Other; p = 0.9878, Mixed Models Analysis; Mean Difference (Final Values) = 0.02, 95% CI 2-sided [-2.52 to 2.56] — Mean difference calculated as [Treatment] - Placebo
Statistical Analysis 3: Comparison: Placebo - DINAMOᵀᴹ Mono vs Linagliptin 5 mg - DINAMOᵀᴹ Mono; [analysis description as in outcome 6, analysis 1]; Test type: Other; p = 0.5670, Mixed Models Analysis; Mean Difference (Final Values) = 3.33, 95% CI 2-sided [-9.00 to 15.65] — Mean difference calculated as [Treatment] - Placebo
Statistical Analysis 4: Comparison: Placebo - DINAMOᵀᴹ Mono vs Empagliflozin Pooled (10 mg and 25 mg) - DINAMOᵀᴹ Mono; [analysis description as in outcome 6, analysis 1]; Test type: Other; p = 0.2348, Mixed Models Analysis; Mean Difference (Final Values) = -6.62, 95% CI 2-sided [-18.19 to 4.95] — Mean difference calculated as [Treatment] - Placebo

9. Secondary Outcome: Percentage of Patients Who Achieve HbA1c <6.5% at the End of 26 Weeks
Description: Percentage of patients who achieve HbA1c <6.5% at the end of 26 weeks.
Time Frame: Baseline (Day 1) and week 26.
Population: The modified intention-to-treat set (mITT) included all patients treated with at least 1 dose of trial medication who had a baseline HbA1c measurement. Missing values were regarded as 'failures'.
Measure: Number; unit: Percentage of subjects
Arm/Group | Placebo - DINAMOᵀᴹ | Linagliptin 5 mg - DINAMOᵀᴹ | Empagliflozin Pooled (10 mg and 25 mg) - DINAMOᵀᴹ | Placebo - DINAMOᵀᴹ Mono | Linagliptin 5 mg - DINAMOᵀᴹ Mono | Empagliflozin Pooled (10 mg and 25 mg) - DINAMOᵀᴹ Mono
Number analyzed (Participants) | 53 | 52 | 52 | 5 | 6 | 6
Percentage of subjects | 9.4 | 15.4 | 21.2 | 40.0 | 16.7 | 16.7
Statistical Analysis 1: Comparison: Placebo - DINAMOᵀᴹ vs Linagliptin 5 mg - DINAMOᵀᴹ; The risk difference of active treatments versus placebo was determined and assessed by an exact 2-sided 95% confidence interval. Exact 95% CI by Chan and Zhang. Asymptotic and two-sided Wald test; Test type: Other; p = 0.3536, Wald test; Rate difference (percentage) = 6.0, 95% CI 2-sided [-7.7 to 19.9] — Difference calculated as [Treatment] - Placebo
Statistical Analysis 2: Comparison: Placebo - DINAMOᵀᴹ vs Empagliflozin Pooled (10 mg and 25 mg) - DINAMOᵀᴹ; [analysis description as in outcome 9, analysis 1]; Test type: Other; p = 0.0914, Wald test; Rate difference (percentage) = 11.7, 95% CI 2-sided [-2.4 to 26.3] — Difference calculated as [Treatment] - Placebo
Statistical Analysis 3: Comparison: Placebo - DINAMOᵀᴹ Mono vs Linagliptin 5 mg - DINAMOᵀᴹ Mono; The risk difference of active treatments versus placebo was determined and assessed by an exact 2-sided 95% confidence interval. Exact 95% CI by Chan and Zhang. Asymptotic and Fisher's exact test; Test type: Other; p = 0.5455, Fisher Exact; Rate difference (percentage) = -23.3, 90% CI 2-sided [-67.9 to 27.1] — Difference calculated as [Treatment] - Placebo
Statistical Analysis 4: Comparison: Placebo - DINAMOᵀᴹ Mono vs Empagliflozin Pooled (10 mg and 25 mg) - DINAMOᵀᴹ Mono; [analysis description as in outcome 9, analysis 3]; Test type: Other; p = 0.5455, Fisher Exact; Rate difference (percentage) = -23.3, 90% CI 2-sided [-67.9 to 27.1] — Difference calculated as [Treatment] - Placebo

10. Secondary Outcome: Percentage of Patients Who Achieve HbA1c <7.0% at the End of 26 Weeks
Description: Percentage of patients who achieve HbA1c <7.0% at the end of 26 weeks.
Time Frame: Baseline (Day 1) and week 26.
Population: as for outcome 9
Measure: Number; unit: Percentage of subjects
Arm/Group | Placebo - DINAMOᵀᴹ | Linagliptin 5 mg - DINAMOᵀᴹ | Empagliflozin Pooled (10 mg and 25 mg) - DINAMOᵀᴹ | Placebo - DINAMOᵀᴹ Mono | Linagliptin 5 mg - DINAMOᵀᴹ Mono | Empagliflozin Pooled (10 mg and 25 mg) - DINAMOᵀᴹ Mono
Number analyzed (Participants) | 53 | 52 | 52 | 5 | 6 | 6
Percentage of subjects | 24.5 | 26.9 | 34.6 | 40.0 | 16.7 | 66.7
Statistical Analysis 1: Comparison: Placebo - DINAMOᵀᴹ vs Linagliptin 5 mg - DINAMOᵀᴹ; [analysis description as in outcome 9, analysis 1]; Test type: Other; p = 0.7789, Wald test; Rate difference (percentage) = 2.4, 95% CI 2-sided [-15.2 to 19.5] — Difference calculated as [Treatment] - Placebo
Statistical Analysis 2: Comparison: Placebo - DINAMOᵀᴹ vs Empagliflozin Pooled (10 mg and 25 mg) - DINAMOᵀᴹ; [analysis description as in outcome 9, analysis 1]; Test type: Other; p = 0.2548, Wald test; Rate difference (percentage) = 10.1, 95% CI 2-sided [-7.7 to 28.1] — Difference calculated as [Treatment] - Placebo
Statistical Analysis 3: Comparison: Placebo - DINAMOᵀᴹ Mono vs Linagliptin 5 mg - DINAMOᵀᴹ Mono; [analysis description as in outcome 9, analysis 3]; Test type: Other; p = 0.5455, Fisher Exact; Rate difference (percentage) = -23.3, 90% CI 2-sided [-67.9 to 27.1] — Difference calculated as [Treatment] - Placebo
Statistical Analysis 4: Comparison: Placebo - DINAMOᵀᴹ Mono vs Empagliflozin Pooled (10 mg and 25 mg) - DINAMOᵀᴹ Mono; [analysis description as in outcome 9, analysis 3]; Test type: Other; p = 0.5671, Fisher Exact; Rate difference (percentage) = 26.7, 90% CI 2-sided [-30.8 to 70.8] — Difference calculated as [Treatment] - Placebo

ADVERSE EVENTS:
Time Frame: Date of first study drug intake until date of last active study drug intake + residual effect period (7 days), up to 402 days.
Description: The treated set (TS) included all patients treated with at least 1 dose of randomised trial medication.
Groups:
- Placebo Pooled - DINAMOᵀᴹ & DINAMOᵀᴹ Mono: Patients from either DINAMOᵀᴹ or DINAMOᵀᴹ Mono randomized to Placebo.
- Linagliptin 5 mg Pooled - DINAMOᵀᴹ & DINAMOᵀᴹ Mono: Patients from either DINAMOᵀᴹ or DINAMOᵀᴹ Mono who either started on Linagliptin or who switched to Linagliptin from Placebo at week 26. 1 film-coated tablet of 5 milligram (mg) Linagliptin once daily.
- Empagliflozin 10 mg Pooled - DINAMOᵀᴹ & DINAMOᵀᴹ Mono: Patients from either DINAMOᵀᴹ or DINAMOᵀᴹ Mono who either started on 10 mg Empagliflozin or switched to 10 mg Empagliflozin from Placebo at week 26. 1 film-coated tablet of 10 milligram (mg) Empagliflozin once daily.
- Empagliflozin 25 mg Pooled - DINAMOᵀᴹ & DINAMOᵀᴹ Mono: Patients from either DINAMOᵀᴹ or DINAMOᵀᴹ Mono who were on Placebo and switched to 25 mg Empagliflozin following re-randomisation at week 26 or who were on 10 mg Empagliflozin and switched to 25 mg Empagliflozin following re-randomisation at week 14. 1 film-coated tablet of 25 mg empagliflozin, taken once daily, until end of treatment.
Arm/Group | Placebo Pooled - DINAMOᵀᴹ & DINAMOᵀᴹ Mono | Linagliptin 5 mg Pooled - DINAMOᵀᴹ & DINAMOᵀᴹ Mono | Empagliflozin 10 mg Pooled - DINAMOᵀᴹ & DINAMOᵀᴹ Mono | Empagliflozin 25 mg Pooled - DINAMOᵀᴹ & DINAMOᵀᴹ Mono
All-Cause Mortality (participants affected / at risk) | 0/58 | 0/77 | 0/74 | 0/29
Serious Adverse Events (participants affected / at risk) | 2/58 | 8/77 | 4/74 | 0/29
Other Adverse Events (participants affected / at risk) | 30/58 | 45/77 | 47/74 | 14/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Pooled - DINAMOᵀᴹ & DINAMOᵀᴹ Mono (N=58) | Linagliptin 5 mg Pooled - DINAMOᵀᴹ & DINAMOᵀᴹ Mono (N=77) | Empagliflozin 10 mg Pooled - DINAMOᵀᴹ & DINAMOᵀᴹ Mono (N=74) | Empagliflozin 25 mg Pooled - DINAMOᵀᴹ & DINAMOᵀᴹ Mono (N=29)
Splenic vein thrombosis (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Systemic inflammatory response syndrome (General disorders) | 1 | 0 | 0 | 0
Breast abscess (Infections and infestations) | 0 | 1 | 0 | 0
Chorioretinitis (Infections and infestations) | 0 | 1 | 0 | 0
Skin candida (Infections and infestations) | 0 | 0 | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Blood glucose increased (Investigations) | 0 | 1 | 0 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 2 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 0 | 0
Tubulointerstitial nephritis (Renal and urinary disorders) | 0 | 0 | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Hypovolaemic shock (Vascular disorders) | 1 | 0 | 0 | 0
Peripheral ischaemia (Vascular disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Pooled - DINAMOᵀᴹ & DINAMOᵀᴹ Mono (N=58) | Linagliptin 5 mg Pooled - DINAMOᵀᴹ & DINAMOᵀᴹ Mono (N=77) | Empagliflozin 10 mg Pooled - DINAMOᵀᴹ & DINAMOᵀᴹ Mono (N=74) | Empagliflozin 25 mg Pooled - DINAMOᵀᴹ & DINAMOᵀᴹ Mono (N=29)
Abdominal pain (Gastrointestinal disorders) | 4 | 5 | 4 | 1
Abdominal pain upper (Gastrointestinal disorders) | 2 | 2 | 2 | 2
Diarrhoea (Gastrointestinal disorders) | 5 | 7 | 3 | 2
Nausea (Gastrointestinal disorders) | 3 | 4 | 3 | 0
Vomiting (Gastrointestinal disorders) | 2 | 8 | 5 | 2
Seasonal allergy (Immune system disorders) | 0 | 0 | 4 | 0
Influenza (Infections and infestations) | 0 | 4 | 3 | 0
Nasopharyngitis (Infections and infestations) | 3 | 6 | 3 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 3 | 5 | 1
Urinary tract infection (Infections and infestations) | 1 | 1 | 5 | 2
Blood ketone body increased (Investigations) | 2 | 8 | 5 | 3
Urine albumin/creatinine ratio increased (Investigations) | 2 | 5 | 1 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 5 | 3 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 7 | 16 | 12 | 5
Vitamin D deficiency (Metabolism and nutrition disorders) | 8 | 6 | 10 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 4 | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 4 | 4 | 0
Dizziness (Nervous system disorders) | 3 | 1 | 4 | 0
Headache (Nervous system disorders) | 9 | 12 | 12 | 3
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 2 | 6 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 6 | 4 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 5 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2022-05-23): https://cdn.clinicaltrials.gov/large-docs/43/NCT03429543/Prot_000.pdf
  • Statistical Analysis Plan (2022-07-28): https://cdn.clinicaltrials.gov/large-docs/43/NCT03429543/SAP_001.pdf